CLINICAL TRIAL: NCT00898365
Title: Renal Tumors Classification, Biology, and Banking Study
Brief Title: Study of Kidney Tumors in Younger Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN03B2; NCI-2009-00416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AREN03B2; CDR0000459797; AREN03B2 (Other: Children's Oncology Group); AREN03B2 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH); UG1CA189958 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2024-08

CONDITIONS: Adult Cystic Nephroma; Anaplastic Kidney Wilms Tumor; Angiolipoma; Cellular Congenital Mesoblastic Nephroma; Classic Congenital Mesoblastic Nephroma; Clear Cell Sarcoma of the Kidney; Congenital Mesoblastic Nephroma; Cystic Partially Differentiated Kidney Nephroblastoma; Diffuse Hyperplastic Perilobar Nephroblastomatosis; Extrarenal Rhabdoid Tumor; Kidney Medullary Carcinoma; Kidney Neoplasm; Kidney Oncocytoma; Kidney Wilms Tumor; Metanephric Adenofibroma; Metanephric Adenoma; Metanephric Stromal Tumor; Metanephric Tumor; Mixed Congenital Mesoblastic Nephroma; Ossifying Renal Tumor of Infancy; Papillary Renal Cell Carcinoma; Renal Cell Carcinoma; Renal Cell Carcinoma Associated With Xp11.2 Translocations/TFE3 Gene Fusions; Rhabdoid Tumor of the Kidney; Wilms Tumor
MeSH Terms: conditions — Angiolipoma; Nephroma, Mesoblastic; Kidney Neoplasms; Oncocytoma, renal; Wilms Tumor; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor, blood, and urine samples

GROUPS / COHORTS (1):
- Ancillary-correlative (renal tumor classification, biology): Tumor tissue, blood, and urine samples are collected for research studies, including immunohistochemistry. CT scans and MRIs are also performed. Loss of heterozygosity analyses (chromosome 1p and 16q) are performed by extraction of DNA. DNA polymorphisms are assayed by polymerase chain reaction using standard methodology. Leftover specimens are archived for future studies. (LOH and INI1 testing discontinued as of April 2014)
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies kidney tumors in younger patients. Collecting and storing samples of tumor tissue, blood, and urine from patients with cancer to study in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Classify patients with renal tumors by histological categorization, surgico-pathological stage, presence of metastases, age at diagnosis, tumor weight, and loss of heterozygosity for chromosomes 1p and 16q, to define eligibility for a series of therapeutic studies.

(As of Amendment 8, this aim is limited to patients with institutionally classified Stage I to IV focal or diffuse anaplasia identified at initial biopsy or primary nephrectomy OR at delayed nephrectomy/second biopsy.)

II. To maintain a biological samples bank to make specimens available to scientists to evaluate additional potential biological prognostic variables and for the conduct of other research by scientists.

SECONDARY OBJECTIVES:

I. To monitor outcome for those patients who are not eligible for a subsequent therapeutic study.

II. To describe whether the pulmonary tumor burden correlates with outcome in Stage IV patients.(Completed as of Amendment 7)

III. To describe the sensitivity and specificity of abdominal computed tomography (CT) by comparison with surgical and pathologic findings for identification of local tumor spread beyond the renal capsule to adjacent muscle and organs, lymph node involvement at the renal hilum and in the retroperitoneum, preoperative tumor rupture and metastases to the liver. (Completed as of Amendment 7)

IV. To compare the sensitivity and specificity of preoperative abdominal CT and MRI for the identification and differentiation of nephrogenic rests and Wilms tumor in children with multiple renal lesions. (Completed as of Amendment 7)

V. To correlate the method of conception (natural versus assisted reproductive technology) with the development of Wilms tumor. (Completed as of Amendment 7)

VI. To evaluate the frequency of integrase interactor 1 (INI1) mutations in renal and extrarenal malignant rhabdoid tumor of the kidney and to determine the incidence of germline and inherited versus somatic mutations to facilitate clinical correlations on the companion study AREN0321. (Completed as of Amendment 7)

OUTLINE:

Tumor tissue, blood, and urine samples are collected for research studies, including immunohistochemistry. CT scans and MRIs are also performed. Loss of heterozygosity analyses (chromosome 1p and 16q) are performed by extraction of DNA. DNA polymorphisms are assayed by polymerase chain reaction using standard methodology. Leftover specimens are archived for future studies. (LOH and INI1 testing discontinued as of April 2014)

Patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the first occurrence of any tumor of the kidney identified on CT scan or MRI are eligible for this study; histologic diagnosis is not required prior to enrollment but is required for all patients once on study
* Eligible tumors include (but are not limited to):

  * Nephroblastic tumors

    * Nephroblastoma (Wilms' tumor) (favorable histology, anaplasia [diffuse, focal])
    * Nephrogenic rests and nephroblastomatosis
    * Cystic nephroma and cystic partially differentiated nephroblastoma
    * Metanephric tumors (metanephric adenoma, metanephric adenofibroma, metanephric stromal tumor)
  * Mesoblastic nephroma (cellular, classic, mixed)
  * Clear cell sarcoma
  * Rhabdoid tumor (any malignant rhabdoid tumor occurring outside the central nervous system [CNS])
  * Renal epithelioid tumors of childhood (papillary renal cell carcinoma, medullary renal cell carcinoma, renal tumors associated with Xp11.2 translocations, oncocytic renal neoplasms after neuroblastoma)
  * Angiolipoma
  * Ossifying renal tumor of infancy
* Patients with the first occurrence of the following tumors are also eligible:

  * Extrarenal nephroblastoma or extrarenal neprogenic rests
  * Malignant rhabdoid tumor occurring anywhere outside the central nervous system
* Required specimens, reports, forms, and copies of imaging studies must be available or will become available for submission and the institution must intend on submitting them as described in the protocol procedures
* For ALL patients, (with exception of bilateral, bilaterally predisposed, multicentric, or unilateral tumor in solitary kidney planning to enroll without biopsy***), the following submissions are required:

  * A complete set of recut hematoxylin and eosin (H & E) slides (including from sampled lymph nodes, if patient had upfront nephrectomy)

    * * Tissue must be from diagnosis, prior to any renal tumor directed chemotherapy or radiation (only exception is for presumed favorable histology Wilms tumor [FHWT] patients discovered to have diffuse anaplastic Wilms tumor [DAWT] at delayed nephrectomy and plan to enroll at delayed nephrectomy)
  * Representative formalin-fixed paraffin-embedded tissue block or if a block is unavailable, 10 unstained slides from a representative block of tumor, if available.

    * Tissue must be from diagnosis, prior to any renal tumor directed chemotherapy or radiation (only exception is for presumed FHWT patients discovered to have DAWT at delayed nephrectomy and plan to enroll at delayed nephrectomy)
  * Institutional pathology report, Specimen Transmittal Form, and Pre-Treatment Pathology Checklist
  * Copies of images and institutional reports of CT and/or MRI abdomen and pelvis, and Pre Treatment Imaging Checklist
  * Copies of images and institutional report of chest CT for all malignant tumors
  * Institutional surgical report(s) and Pre-Treatment Surgical Checklist
  * CRFs: Staging Checklist and Metastatic Disease Form (if metastatic disease is noted on imaging)

    * Patients with bilateral, bilaterally predisposed, multicentric, or unilateral tumor in solitary kidney planning to enroll without biopsy via imaging only - these patients will not have central review or have a risk assignment issued, but may contribute to specimen banking for future research. However, if biopsy is done, tissue must be submitted as for other renal tumors, and initial risk assignment will require pathology and surgical rapid central reviews. The Specimen Transmittal Form and Pre Treatment Pathology Checklist are also needed.
  * Please note: if the above required items are not received within 120 days of study enrollment, the patient will be considered off study
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients newly diagnosed with kidney tumors
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2006-02-27 (Actual); Primary Completion 2100-01-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Up to 5 years from study enrollment
  Time from diagnosis to the earliest occurrence of disease progression (if enrolling with measurable disease), first relapse (if enrolling without measurable disease), secondary malignancy, or death. Analysis plans are specific to individual COG-approved projects and biology protocols.
Overall survival | Up to 5 years from study enrollment
  Time from diagnosis to death. Analysis plans are specific to individual COG-approved projects and biology protocols.

SECONDARY OUTCOMES:
Loss of heterozygosity (LOH testing discontinued as of April 2014) | Baseline
  Evaluation of LOH (1p and 16q) status was performed in select patients with newly diagnosed favorable histology Wilms Tumor during the time that AREN0532 and AREN0533 were open to enrollment, in order to direct patients to the appropriate therapeutic protocol and study arm as well as validate the markers' prognostic value.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Mullen, Principal Investigator — Children's Oncology Group
Locations (248):
- United States (214):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Cabell-Huntington Hospital, Huntington, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (11):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- Schneider Children's Medical Center of Israel, Petah Tikua, Israel
- New Zealand (3):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Children's Hospital, Wellington
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- Swiss Pediatric Oncology Group - Bern, Bern, Switzerland

REFERENCES:
- [Derived] Benedetti DJ, Renfro LA, Tfirn I, Daw NC, Kalapurakal JA, Ehrlich PF, Khanna G, Perlman E, Warwick A, Gow KW, Paulino AC, Seibel NL, Grundy P, Fernandez CV, Geller JI, Mullen EA, Dome JS. Treatment and outcomes of clear cell sarcoma of the kidney: A report from the Children's Oncology Group studies AREN0321 and AREN03B2. Cancer. 2024 Jul 1;130(13):2361-2371. doi: 10.1002/cncr.35266. Epub 2024 Feb 23. PMID 38396300
- [Derived] Benedetti DJ, Varela CR, Renfro LA, Tornwall B, Dix DB, Ehrlich PF, Glick RD, Kalapurakal J, Perlman E, Gratias E, Seibel NL, Geller JI, Khanna G, Malogolowkin M, Grundy P, Fernandez CV, Dome JS, Mullen EA. Treatment of children with favorable histology Wilms tumor with extrapulmonary metastases: A report from the COG studies AREN0533 and AREN03B2 and NWTSG study NWTS-5. Cancer. 2024 Mar 15;130(6):947-961. doi: 10.1002/cncr.35099. Epub 2023 Nov 7. PMID 37933882
- [Derived] Parsons LN, Mullen EA, Geller JI, Chi YY, Khanna G, Glick RD, Aldrink JH, Vallance KL, Kim Y, Fernandez CV, Dome JS, Perlman EJ. Outcome analysis of stage I epithelial-predominant favorable-histology Wilms tumors: A report from Children's Oncology Group study AREN03B2. Cancer. 2020 Jun 15;126(12):2866-2871. doi: 10.1002/cncr.32855. Epub 2020 Apr 8. PMID 32267967